CLINICAL TRIAL: NCT03702270
Title: The Effect of Providing Stratification of Low Risk Penicillin Allergies on Penicillin Allergy Label Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cosby Stone, Instructor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 181734
Record Dates: First submitted 2018-10-08; First posted 2018-10-11 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Penicillin Allergy

STUDY DESIGN:
Intervention Model Description: During the trial, randomization will occur using a stepped wedge cluster randomized controlled trial design. Medical units at VUMC will be assigned to clusters. A single cluster will be selected for intervention at the outset of the trial. Subsequent additional clusters will first contribute to the control group, and be selected to randomly cross over to the intervention group at regular intervals of 1 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penicillin Allergic Floor Patients- Experimental (Experimental): The intervention will provide access to a best-practices alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  Interventions: Other: Penicillin Allergic Risk Stratification Best Practice Alert
- Penicillin Allergic Floor Patients- Control (No Intervention): Patients will receive current standard of care for penicillin allergy, which typically involves physician judgement on challenges versus consultation of allergy service.

INTERVENTIONS:
Other: Penicillin Allergic Risk Stratification Best Practice Alert — Providing best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  Arms: Penicillin Allergic Floor Patients- Experimental

SUMMARY:
Currently it is estimated that at least 25 million people in the United States are labeled as penicillin allergic although less than 1.5 million of these are truly allergic. Although combined skin testing and oral challenge is an evidence-based de-labeling strategy the high burden of penicillin allergy labels means these services are available only through specialty allergy practices. There is therefore a need to provide evidence for alternative penicillin de-labeling strategies such as direct oral challenge. Previous studies have utilized quasi-experimental designs. Test dose challenges are currently recommended as a strategy for removal of low risk drug allergies, but the current experience is limited to single arm observational studies and evidence-based strategies for identifying low risk patients are lacking. Our objective is to demonstrate the benefit of providing risk stratification in removing penicillin allergy labels for low risk penicillin allergy patients in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* VUMC patients age 18 or older with a penicillin allergy reported in their chart, and are medically stable, currently admitted to stepdown unit or regular floor bed.

Exclusion Criteria:

* Patients with a penicillin allergy reported in their chart, but who are currently medically unstable.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2052 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cosby Stone, MD, MPH, Principal Investigator — Vanderbilt University Medical Center; Chris Lindsell, PhD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Control Group: Patients who did not have 24-hour exposure to a study unit where the intervention was active but did have at least 24-hour exposure to a control unit. Intervention Group: Patients who had a 24-hour exposure to a study unit at any time where the intervention was active. Patients could move through different hospital units throughout the course of clinical care. The number of participants per sequence reflects the first unit where a participant had a 24-hour exposure.
Units Other Than Participants: Medical Units
Groups:
- Sequence A: 1 month control, then 12 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence B: 2 months control, then 11 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence C: 3 month control, then 10 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence D: 4 months control, then 9 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence E: 5 months control, then 8 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence F: 6 months control, then 7 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence G: 7 months control, then 6 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence H: 8 months control, then 5 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence I: 9 months control, then 4 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence J: 10 months control, then 3 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence K: 11 months control, then 2 months of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
- Sequence L: 12 months control, then 1 month of intervention. The intervention will provide access to a best-practice alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  The penicillin allergic risk stratification Best Practice Alert provides best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
  In this stepped wedge design, all units have a period of being in control, and then providing the intervention. Medical units transitioned from the control condition to the intervention condition at monthly intervals. Units remained in the intervention condition once transitioned.
Period: Control
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F | Sequence G | Sequence H | Sequence I | Sequence J | Sequence K | Sequence L
Started | 17; 1 Medical Units | 31; 1 Medical Units | 51; 1 Medical Units | 27; 1 Medical Units | 53; 1 Medical Units | 65; 1 Medical Units | 97; 1 Medical Units | 87; 1 Medical Units | 125; 1 Medical Units | 179; 1 Medical Units | 191; 1 Medical Units | 111; 1 Medical Units
Completed | 17; 1 Medical Units | 31; 1 Medical Units | 51; 1 Medical Units | 27; 1 Medical Units | 53; 1 Medical Units | 65; 1 Medical Units | 97; 1 Medical Units | 87; 1 Medical Units | 125; 1 Medical Units | 179; 1 Medical Units | 191; 1 Medical Units | 111; 1 Medical Units
Not Completed | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units
Period: Intervention
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F | Sequence G | Sequence H | Sequence I | Sequence J | Sequence K | Sequence L
Started | 237; 1 Medical Units | 138; 1 Medical Units | 113; 1 Medical Units | 65; 1 Medical Units | 76; 1 Medical Units | 70; 1 Medical Units | 77; 1 Medical Units | 62; 1 Medical Units | 61; 1 Medical Units | 59; 1 Medical Units | 41; 1 Medical Units | 19; 1 Medical Units
Completed | 237; 1 Medical Units | 138; 1 Medical Units | 113; 1 Medical Units | 65; 1 Medical Units | 76; 1 Medical Units | 70; 1 Medical Units | 77; 1 Medical Units | 62; 1 Medical Units | 61; 1 Medical Units | 59; 1 Medical Units | 41; 1 Medical Units | 19; 1 Medical Units
Not Completed | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units | 0; 0 Medical Units

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Penicillin Allergic Floor Patients- Experimental | Penicillin Allergic Floor Patients- Control | Total
Number analyzed (Participants) | 1018 | 1034 | 2052
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.6 [51.0 to 73.7] | 61.7 [50.0 to 72.6] | 63.1 [50.3 to 73.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 596 | 593 | 1189
  Male | 422 | 441 | 863
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 8 | 2 | 10
  Race: More Than One Race | 8 | 10 | 18
  Race: Asian | 1 | 4 | 5
  Race: Black or African American | 165 | 156 | 321
  Race: Unknown/Not Reported | 9 | 15 | 24
  Race: White | 827 | 847 | 1674
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic, Latino | 448 | 445 | 893
  Ethnicity: Hispanic, Latino | 14 | 19 | 33
  Ethnicity: Unknown/Not Reported | 556 | 570 | 1126
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1018 | 1034 | 2052

OUTCOME MEASURES:

1. Primary Outcome: Penicillin Allergy Label Removal
Description: The percentage of patients with low risk penicillin allergy whose labels are removed from the medical chart's allergy section.
Time Frame: Hospital discharge at approximately 4 days after admission
Measure: Count of Participants; unit: Participants
Arm/Group | Penicillin Allergic Floor Patients- Experimental | Penicillin Allergic Floor Patients- Control
Number analyzed (Participants) | 1018 | 1034
Participants | 45 | 31

2. Secondary Outcome: Adverse Events (in Particular, Reported Allergic Events)
Description: The percentage of penicillin allergic patients challenged with amoxicillin who reported adverse events
Time Frame: Hospital discharge at approximately 4 days after admission
Measure: Count of Participants; unit: Participants
Groups:
- Penicillin Allergic Floor Patients Who Received Amoxicillin Challenge - Experimental: Patients in the intervention group who received an amoxicillin challenge.
  The intervention will provide access to a best-practices alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  Penicillin Allergic Risk Stratification Best Practice Alert: Providing best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
- Penicillin Allergic Floor Patients Who Received Amoxicillin Challenge - Control: Patients in the control group who received an amoxicillin challenge.
  Patients will receive current standard of care for penicillin allergy, which typically involves physician judgement on challenges versus consultation of allergy service.
Arm/Group | Penicillin Allergic Floor Patients Who Received Amoxicillin Challenge - Experimental | Penicillin Allergic Floor Patients Who Received Amoxicillin Challenge - Control
Number analyzed (Participants) | 27 | 21
Participants | 0 | 0

3. Secondary Outcome: Communication About Penicillin Allergy in Discharge Summary
Description: The percentage of penicillin allergic patients whose discharge summary contains information about penicillin allergy at discharge.
Time Frame: Hospital discharge at approximately 4 days after admission
Measure: Count of Participants; unit: Participants
Groups:
- Patient Communication About Allergy Label Removal- Experimental: Penicillin allergic floor patients in the intervention group who received an amoxicillin challenge, had their allergy label removed, and received discharge communication.
  The intervention will provide access to a best-practices alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  Penicillin Allergic Risk Stratification Best Practice Alert: Providing best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
- Patient Communication About Allergy Label Removal- Control: Penicillin allergic floor patients in the control group who received amoxicillin challenge, had their allergy label removed, and received discharge communication.
  Patients will receive current standard of care for penicillin allergy, which typically involves physician judgement on challenges versus consultation of allergy service.
Arm/Group | Patient Communication About Allergy Label Removal- Experimental | Patient Communication About Allergy Label Removal- Control
Number analyzed (Participants) | 26 | 20
Participants
  Yes | 21 | 14
  No | 5 | 2
  Missing | 0 | 4

4. Secondary Outcome: Antibiotic Utilization by Patients
Description: The number of changes or new starts of penicillin or cephalosporin treatments as a result of penicillin allergy label removal and the proportion of patients experiencing this event, this will be looked at as "Same hospitalization" as the challenge or "Subsequent Utilization"
Time Frame: Hospital discharge at approximately 4 days after admission and from 3-18 months of follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Penicillin Allergic Floor Patients- Experimental | Penicillin Allergic Floor Patients- Control
Number analyzed (Participants) | 1018 | 1034
Participants
  Same Hospitalization: Never | 680 | 715
  Same Hospitalization: Ever | 338 | 319
  3 Months Post-Randomization: Never | 826 | 847
  3 Months Post-Randomization: Ever | 192 | 187
  18 Months Post-Randomization: Never | 602 | 627
  18 Months Post-Randomization: Ever | 416 | 407

5. Secondary Outcome: Durability of Penicillin Allergy Label Removal
Description: The percentage of penicillin allergic patients whose penicillin allergy labels were removed at discharge whose labels are not reentered into the chart.
Time Frame: Hospital discharge at approximately 4 days after admission and from 3-18 months of follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Penicillin Allergic Floor Patients- Experimental | Penicillin Allergic Floor Patients- Control
Number analyzed (Participants) | 45 | 31
Participants
  3 Months Post-Randomization | 44 | 28
  18 Months Post-Randomization | 43 | 29

6. Secondary Outcome: Receipt of Risk Stratification Tool Assessment
Description: Number of patients with a penicillin allergy label who received a risk assessment.
Time Frame: Hospital discharge at approximately 4 days after admission
Measure: Count of Participants; unit: Participants
Arm/Group | Penicillin Allergic Floor Patients- Experimental | Penicillin Allergic Floor Patients- Control
Number analyzed (Participants) | 1018 | 1034
Participants | 86 | 27

7. Secondary Outcome: Time to Penicillin Allergy Label Return
Description: For those patients who underwent a penicillin allergy label removal and it returns, we will compare the date the allergy label returned with the date it was removed
Time Frame: From 3-18 months of follow up
Population: Intervention arm had 40 patients whose labels did not return. The control had 27 patients whose labels did not return.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Time to Penicillin Allergy Label Return - Experimental: Penicillin allergic floor patients in the intervention group who received an amoxicillin challenge and had their allergy label removed.
  The intervention will provide access to a best-practices alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  Penicillin Allergic Risk Stratification Best Practice Alert: Providing best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.
- Time to Penicillin Allergy Label Return - Control: Penicillin allergic floor patients in the control group who received amoxicillin challenge and had their allergy label removed.
  Patients will receive current standard of care for penicillin allergy, which typically involves physician judgement on challenges versus consultation of allergy service.
Arm/Group | Time to Penicillin Allergy Label Return - Experimental | Time to Penicillin Allergy Label Return - Control
Number analyzed (Participants) | 5 | 4
days | 35.62 [22.01 to 115.91] | 52.89 [36.49 to 109.98]

8. Secondary Outcome: Penicillin Utilization by Patients
Description: The number of changes or new starts of penicillin treatments as a result of penicillin allergy label removal and the proportion of patients experiencing this event, this will be looked at as "Same hospitalization" as the challenge or "Subsequent Utilization"
Time Frame: Hospital discharge at approximately 4 days after admission and from 3-18 months of follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Penicillin Allergic Floor Patients- Experimental | Penicillin Allergic Floor Patients- Control
Number analyzed (Participants) | 1018 | 1034
Participants
  Same Hospitalization | 84 | 57
  3 Months Post-Randomization | 68 | 46
  18 Months Post-Randomization | 173 | 140

9. Secondary Outcome: Cephalosporin Utilization by Patients
Description: The number of changes or new starts of cephalosporin treatments as a result of penicillin allergy label removal and the proportion of patients experiencing this event, this will be looked at as "Same hospitalization" as the challenge or "Subsequent Utilization"
Time Frame: Hospital discharge at approximately 4 days after admission and from 3-18 months of follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Penicillin Allergic Floor Patients- Experimental | Penicillin Allergic Floor Patients- Control
Number analyzed (Participants) | 1018 | 1034
Participants
  Same Hospitalization | 293 | 297
  3 Months Post-Randomization | 156 | 173
  18 Months Post-Randomization | 363 | 379

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the index hospitalization, from randomization to discharge (~4 days post-randomization).
Arm/Group | Penicillin Allergic Floor Patients- Experimental | Penicillin Allergic Floor Patients- Control
All-Cause Mortality (participants affected / at risk) | 0/1018 | 0/1034
Serious Adverse Events (participants affected / at risk) | 0/1018 | 0/1034
Other Adverse Events (participants affected / at risk) | 0/1018 | 0/1034

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT03702270/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03702270/SAP_002.pdf